CLINICAL TRIAL: NCT06000449
Title: Center M: Digital Health Innovation Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ellen Tilden, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00026642; 1R41MH134692 (NIH)
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Perinatal Depression
Keywords: Maternal Mental Health; Telehealth
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Center M (Experimental): This intervention will include digital PD screening as well as four weekly one-hour group telehealth Mindfulness Cognitive Behavioral Therapy sessions and digitally delivered home practice materials for skill building between online group sessions.
  Interventions: Behavioral: Center M
- Treatment as Usual (TAU) (Active Comparator): This arm will receive the current standard of care, which includes a paper-based PD screening and a PD educational handout.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Center M — Digital mental health platform. Screening and prevention activities will be provided through the Center M platform, telehealth group mindfulness sessions, and digitally delivered home practice materials.
  Arms: Center M
Behavioral: Treatment as Usual — Paper screening and PD handout.
  Arms: Treatment as Usual (TAU)

SUMMARY:
Center M is a digital health solution to Perinatal Depression (PD) which provides an alternative to Mindfulness Based Cognitive Therapy - Perinatal Depression (MBCT-PD). Center M shifts treatment to a telehealth model, reduces the number of sessions, and transitions home practice materials to a digital format. This study will include a clinical trial in which participants will be randomized to the Center M treatment with smartphone app delivery of homework compared to treatment as usual (TAU).

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant
* Age 18-50 years
* Fluent in English
* Available and able to attend online group scheduled meetings

Exclusion Criteria:

* Current or past enrollment in a mindfulness-based intervention group

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Screening Rate | 6 weeks postpartum
  Rates of PD screening in Center M and TAU groups.
PD Symptoms at baseline | Initial screening pre-intervention
  PD symptom severity measured by two validated depression screening instruments, The Center for Epidemiologic Studies Depression - Revised (CESD-R) and The Edinburgh Postnatal Depression Scale (EPDS).
PD Symptoms post intervention | Two weeks post intervention
  PD symptom severity measured by two validated depression screening instruments, The Center for Epidemiologic Studies Depression - Revised (CESD-R) and The Edinburgh Postnatal Depression Scale (EPDS).
PD Symptoms post intervention | Four weeks post intervention
  PD symptom severity measured by two validated depression screening instruments, The Center for Epidemiologic Studies Depression - Revised (CESD-R) and The Edinburgh Postnatal Depression Scale (EPDS).
PD Symptoms postpartum | Six weeks postpartum
  PD symptom severity measured by two validated depression screening instruments, The Center for Epidemiologic Studies Depression - Revised (CESD-R) and The Edinburgh Postnatal Depression Scale (EPDS).

SECONDARY OUTCOMES:
Participant Satisfaction | Six weeks postpartum
  Participant satisfaction with PD care measured by The Client Satisfaction Questionnaire - 8 (CSQ-8).

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Tilden, PhD, CNM, FACNM, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with IRB #17203 (MBCT-PD Feasibility) #19166 (The Roo Study on Mom and Baby Well-Being) #18579 (Prenatal Environment and Child Health), #19004 (Maternal Well-Being Study) or #20186 (Parents Engaging Infants Study or PENGuIN). This is included in the consent form. Data will be linked between studies using non-HIPAA based participant identification numbers. Any research staff transferring data will be included on all of the study IRB protocols.
Access Criteria: Data for specific participants who need to be linked across studies will be deidentified and transferred. Data is only accessible on an individual user basis by Principal Investigators. Any research staff transferring data will be included on all of the study IRB protocols.